CLINICAL TRIAL: NCT00403507
Title: Physical Activity as a Treatment of Mild-Stage Probable Alzheimer's Disease
Brief Title: Exercise Treatment of Mild-Stage Probable Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other)
Responsible Party: Kelly Davis Garrett, PhD, Intermountain Healthcare
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kelly Garrett
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2006-11

CONDITIONS: Alzheimer Disease; Memory Disorders; Dementia
Keywords: Mild Dementia; Mild Alzheimer; Cognitive Impairment; Cholinesterase Inhibitor; Exercise; Physical activity; Behavior; Memory loss
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Dementia; Cognitive Dysfunction; Motor Activity; Behavior | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clean Control (No Intervention): Probable Alzheimer's disease in the context of no excluding medical conditions.
  Interventions: Behavioral: Participation in a monitored exercise program
- CoMorbid Control (No Intervention): Probable Alzheimer's disease in the context of well-controlled comorbid medical conditions.
  Interventions: Behavioral: Participation in a monitored exercise program
- Clean Exercise (Experimental): Probable Alzheimer's disease in the context no comorbid medical conditions.
  Interventions: Behavioral: Personalized aerobic and strength training.
- CoMorbid Exercise (Experimental): Probable Alzheimer's disease in the context of well-controlled comorbid medical conditions.
  Interventions: Behavioral: Personalized aerobic and strength training.

INTERVENTIONS:
Behavioral: Participation in a monitored exercise program — No contact with control group during 20 weeks.
  Arms: Clean Control; CoMorbid Control
Behavioral: Personalized aerobic and strength training. — Three-days per week for 20 weeks at hospital gym under supervision of exercise specialist.
  Arms: Clean Exercise; CoMorbid Exercise

SUMMARY:
The purpose of the study is to determine if participation in an exercise program helps memory loss from getting worse, and if it improves daily functioning and attitudes of those with probable Alzheimer's disease. It will involve participation of both the person with memory loss and someone who knows their daily activities (e.g., husband, wife, adult child, or caregiver).

DETAILED DESCRIPTION:
Currently, there is no cure for the memory loss associated with Alzheimer's disease, though some medications can help it from getting worse. The research study will help to answer the question if participation in an exercise program helps memory loss from getting worse, and if it improves daily functioning and attitudes of those with probable Alzheimer's disease. It will involve participation of both the person with memory loss and someone who knows their daily activities.

The research study is a randomized-control trial: some participants will be picked to participate in the exercise program, while others will not. Their memory, thinking abilities, activities, and attitudes will be measured at baseline and follow-up assessment 5-6 months later. Participants are in good health, and are treated with a cholinesterase inhibitor for memory loss (standard treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age is 65 through 89 years old.
* Completed more than an 8th grade education.
* Native English speaker.
* Diagnosis of probable Alzheimer's disease by a primary care physician or specialty clinic.
* Taking a cholinesterase inhibitor at a therapeutic dose for at least two weeks prior to admission to study (following minimum titration of four weeks), but no other prescribed medication for cognitive functioning (e.g., memantine/Namenda).
* May have one unstable physical illness that is being treated or a few controlled physical illnesses, is on few medications, and appears no more than mildly ill.
* Treated stable hypertension & hyperlipidemia are permissible, but resting blood pressure must be <170/100 mm Hg.
* Normal TSH & Vitamin B12 levels, as confirmed by laboratory data within 3 years.
* Able to participate a three-day/week physical activity program (No orthopedic, neurologic, or behavioral limitations that may preclude exercise training) for up to 6 months.
* Patient has a knowledgeable informant who can report the day-to-day activities of participant (e.g., spouse, adult child, paid caregiver).
* Able to give assent/consent to research study.

Exclusion Criteria:

* History of learning or developmental disability.
* Treatment with hormone replacement therapy during the last year.
* History of psychiatric condition (including depression).
* Evidence of serious cardiac condition or significant small vessel disease (e.g., heart bypass surgery, angina, arrhythmia, dyspnea, insulin-dependent diabetes with neuropathy, confluent white matter alterations on structural MRI or CT scan).
* History of neurologic condition (e.g., large vessel stroke, seizures, Parkinsonism).
* History of heavy metals exposure.
* History of sleep disturbance (e.g., treated apnea, insomnia).
* History of brain injury (including concussion of >10 minutes).
* History of delirium (change in mental status due to medications) for the past year.
* No pharmaceutical treatment for mood currently, or history of longstanding depression.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
For the intervention group: Change in cognitive performance relative to baseline | baseline & 20 week follow-up
Group differences in cognitive performance following intervention and relative to wait-list control group | baseline & 20 week follow-up
For the intervention group: Change in attitudes, including self-report of well-being and cognitive abilities relative to baseline | baseline & 20 week follow-up
Group differences in attitudes, including self-report of well-being, following intervention and relative to wait-list control group | baseline & 20 week follow-up

SECONDARY OUTCOMES:
For the intervention group: Change in knowledgeable informant's ratings of function, behavior, and attitudes | baseline & 20 week follow-up
Group differences in knowledgeable informant's ratings of function, behavior, and attitudes following intervention and relative to wait-list control group | baseline & 20 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Garrett, Ph.D., Principal Investigator — Intermountain Health Care- LDS Hosptial
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States